CLINICAL TRIAL: NCT05642858
Title: Text Education About Cardiovascular Health and HIV (TEACH-HIV)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22-36653; T32HL007731 (NIH)
Record Dates: First submitted 2022-11-18; First posted 2022-12-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: HIV; Human Immunodeficiency Virus; Cardiovascular Diseases; Atherosclerosis
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Cardiovascular Diseases; Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): The intervention arm will receive education about HIV and heart disease risk via mobile phone text messages for up to 6 months. They will receive the text messages 3-5 times per week. The messages will include information about HIV and risk of heart disease and information about how to reduce heart disease risk. The intervention arm will also receive brief monthly surveys via a digital research platform.
  Interventions: Behavioral: Digital Educational Messaging
- Control Arm (No Intervention): The control arm will not receive the educational text messages. They will receive brief monthly surveys via a digital research platform.

INTERVENTIONS:
Behavioral: Digital Educational Messaging — Education via mobile phone text messages for up to 6 months.
  Arms: Intervention Arm

SUMMARY:
The overall objective is to evaluate the efficacy of educational text messages to reduce cardiovascular risk among persons living with HIV (PLWH).

ELIGIBILITY:
Inclusion Criteria:

* HIV positive
* At least 40 years of age
* English-speaking

Exclusion Criteria:

* Existing clinical atherosclerotic cardiovascular disease (ASCVD)
* Pregnant
* Unwilling/unable to provide informed consent
* Does not own a smartphone

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2023-03-12 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with controlled blood pressure | 6 months
  Proportion of participants with blood pressure < 130/80 mmHg as recorded in the electronic health record (EHR).

SECONDARY OUTCOMES:
Number of cardiovascular risk factors controlled | 6 months
  Total of 8 risk factors: diet, physical activity, nicotine exposure, sleep health, body mass index, blood lipids, blood glucose, blood pressure. Risk factors will be assessed using self-report and EHR data. Risk factor control will be defined based on the American Heart Association's (AHA) Life's Essential 8.
Self-perceived cardiovascular risk | 6 months
  Measured by self-report using questions adapted from the patient and provider assessment of lipid management (PALM) registry.
Systolic blood pressure | 6 months
  Evaluated using EHR data.
Cholesterol | 6 months
  Non-HDL cholesterol, total cholesterol, LDL cholesterol (in mg/dL), as evaluated using EHR data.
Physical activity | 6 months
  Minutes/week, measured via self-report using the International Physical Activity Questionnaire (IPAQ).
Physical activity | 6 months
  Measured via step count.
Mediterranean diet | 6 months
  Measured using the Mediterranean Eating Pattern for Americans (MEPA) tool, as scored by AHA's Life's Essential 8. Score ranges 0-16, with higher scores representing better outcomes.
Proportion of current smokers | 6 months
  Measured via self-report.
Blood sugar control | 6 months
  Evaluated using EHR data on hemoglobin A1c and fasting blood glucose. Blood sugar control will be defined based on the AHA's Life's Essential 8 definitions.
Body mass index | 6 months
  Evaluated in kg/m2 using EHR data.
Proportion of patients on guideline-based therapy | 6 months
  Proportion of patients on anti-hypertensive medications, statins, and aspirin, among those who meet criteria for therapy based on American Heart Association / American College of Cardiology (AHA/ACC) guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Megan McLaughlin, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - University of California San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No